CLINICAL TRIAL: NCT01399164
Title: Cobalamin Absorption From Fortified Food in Older Adults With and Without Proton Pump Inhibitor Induced Achlorhydria
Brief Title: Cobalamin Absorption From Fortified Food
Acronym: FL-72
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WHNRC 242621-1
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Vitamin B-12 Deficiency; Achlorhydria
Keywords: Vitamin B-12
MeSH Terms: conditions — Vitamin B 12 Deficiency; Achlorhydria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fortified Bread (Experimental): A single serving of 14C-B12 fortified bread
  Interventions: Other: 14C-B12 fortified bread

INTERVENTIONS:
Other: 14C-B12 fortified bread — A single serving of 14C-B12 fortified bread

SUMMARY:
To determine B12 bioavailability from 14C-B12 fortified bread in healthy subjects and in subjects with proton pump inhibitor induced achlorhydria.

DETAILED DESCRIPTION:
Cobalamin (vitamin B12) deficiency is highly prevalent in the US and worldwide. Deficiency is most common in the elderly, with an average prevalence ≈25% over age 60 y. About 40% of older persons with low serum cobalamin have food cobalamin malabsorption (F-CM), in which gastric atrophy/achlorhydria and/or dysfunction is implicated. Because of the prevalence of deficiency in those over age 60 y, it is generally recommended that the elderly consume a higher proportion of their cobalamin from fortified foods than what is recommended for younger people. However there is considerable debate about whether crystalline cobalamin is absorbed as well by the elderly with F-CM as it is by younger people, especially if it is added as a fortificant to food. The data to be collected in this study will provide information useful to on-going deliberations concerning the future fortification of wheat flour with vitamin B12 in the United States.

ELIGIBILITY:
Inclusion Criteria:

* good overall health
* normal absorptive capacity (controls) or with a serum B12 <300 pg/mL and a pepsinogen I level >100 μg/L (ACs).
* All subjects must be available to complete the protocol

Exclusion Criteria:

* Any chronic health disorder
* Anemia of any kind
* Renal insufficiency
* excessive alcohol consumption
* Prior GI surgery
* Use of OTC or prescription drugs that interfere with B-12 absorption or metabolism
* Use of vitamin supplements
* Pregnancy or lactation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
B12 bioavailability | 8 Days
  B12 bioavailability from 14C-B12 fortified bread

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Allen, PhD, Principal Investigator — WHNRC, ARS, University of California Davis
Locations (1):
- Western Human Nutrition Center, University of California Davis, Davis, California, United States